CLINICAL TRIAL: NCT03164616
Title: A Phase III, Randomized, Multi-Center, Open-Label, Comparative Global Study to Determine the Efficacy of Durvalumab or Durvalumab and Tremelimumab in Combination With Platinum-Based Chemotherapy for First-Line Treatment in Patients With Metastatic Non Small-Cell Lung Cancer (NSCLC) (POSEIDON)
Brief Title: Study of Durvalumab + Tremelimumab With Chemotherapy or Durvalumab With Chemotherapy or Chemotherapy Alone for Patients With Lung Cancer (POSEIDON).
Acronym: POSEIDON
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D419MC00004; 2017-000920-81 (EudraCT Number)
Record Dates: First submitted 2017-05-22; First posted 2017-05-23 (Actual); Results first posted 2022-04-07 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Non Small Cell Lung Cancer NSCLC
Keywords: NSCLC; Programmed cell death ligand 1 (PD-L1); Durvalumab; Tremelimumab; Progression-free survival (PFS); Overall survival (OS)
MeSH Terms: interventions — durvalumab; tremelimumab; Albumin-Bound Paclitaxel; Carboplatin; Gemcitabine; Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Arm 1 (Experimental): durvalumab + tremelimumab combination therapy + SoC chemotherapy
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Drug: Abraxane + carboplatin; Drug: Gemcitabine + cisplatin; Drug: Gemcitabine + carboplatin; Drug: Pemetrexed + carboplatin; Drug: Pemetrexed + cisplatin
- Treatment Arm 2 (Experimental): durvalumab monotherapy + SoC chemotherapy
  Interventions: Drug: Durvalumab; Drug: Abraxane + carboplatin; Drug: Gemcitabine + cisplatin; Drug: Gemcitabine + carboplatin; Drug: Pemetrexed + carboplatin; Drug: Pemetrexed + cisplatin
- Treatment Arm 3 (Active Comparator): SoC chemotherapy alone
  Interventions: Drug: Abraxane + carboplatin; Drug: Gemcitabine + cisplatin; Drug: Gemcitabine + carboplatin; Drug: Pemetrexed + carboplatin; Drug: Pemetrexed + cisplatin

INTERVENTIONS:
Drug: Durvalumab — IV infusions every 3 weeks for 12 weeks (4 cycles) and every 4 weeks thereafter until disease progression or other discontinuation criteria
  Arms: Treatment Arm 1; Treatment Arm 2
Drug: Tremelimumab — IV infusions every 3 weeks for 12 weeks (4 cycles). An additional dose of tremelimumab will be administered in the week 16.
  Arms: Treatment Arm 1
Drug: Abraxane + carboplatin — Standard of care chemotherapy (squamous and non-squamous patients): Abraxane 100 mg/m2 on Days 1, 8, and 15 of each 21-day cycle. Carboplatin Area under the plasma drug concentration-time curve (AUC) 5 or 6 via IV infusion on Day 1 of each 21-day cycle for 4 to 6 cycles (ie, 4 cycles for Treatment Arms 1 and 2 and 4 to 6 cycles for Treatment Arm 3).
Drug: Gemcitabine + cisplatin — Standard of care chemotherapy (squamous patients only): Gemcitabine 1000 or 1250 mg/m2 via IV infusion on Days 1 and 8 of each 21-day cycle + cisplatin 75 mg/m2 via IV infusion on Day 1 of each 21-day cycle, for 4 to 6 cycles (ie, 4 cycles for Treatment Arms 1 and 2 and 4 to 6 cycles for Treatment Arm 3).
Drug: Gemcitabine + carboplatin — Standard of care chemotherapy (squamous patients only): Gemcitabine 1000 or 1250 mg/m2 via IV infusion on Days 1 and 8 of each 21-day cycle + carboplatin AUC 5 or 6 via IV infusion on Day 1 of each 21-day cycle for 4 to 6 cycles (ie, 4 cycles for Treatment Arms 1 and 2 and 4 to 6 cycles for Treatment Arm 3).
Drug: Pemetrexed + carboplatin — Standard of care chemotherapy (non-squamous patients only): Pemetrexed 500 mg/m2 and carboplatin AUC 5 or 6 via IV infusion on Day 1 of each 21-day cycle for 4 to 6 cycles (ie, 4 cycles for Treatment Arms 1 and 2 and 4 to 6 cycles for Treatment Arm 3); then continue pemetrexed 500 mg/m2 maintenance [i.e., q4w for Treatment Arms 1 and 2. For Treatment Arm 3, Pemetrexed maintenance therapy can be given either q3w or q4w (dependent on Investigator decision and local standards)] until objective disease progression.
Drug: Pemetrexed + cisplatin — Standard of care chemotherapy (non-squamous patients only): Pemetrexed 500 mg/m2 and cisplatin 75 mg/m2 via IV infusion on Day 1 of each 21-day cycle, for 4 to 6 cycles (ie, 4 cycles for Treatment Arms 1 and 2 and 4 to 6 cycles for Treatment Arm 3); then continue pemetrexed 500 mg/m2 maintenance [i.e., q4w for Treatment Arms 1 and 2. For Treatment Arm 3, Pemetrexed maintenance therapy can be given either q3w or q4w (dependent on Investigator decision and local standards)] until objective disease progression.

SUMMARY:
This is a randomized, open-label, multi-center, global, Phase III study to determine the efficacy and safety of durvalumab + tremelimumab combination therapy + Standard of care (SoC) chemotherapy or durvalumab monotherapy + SoC chemotherapy versus SoC chemotherapy alone as first line treatment in patients with metastatic non small-cell lung cancer (NSCLC) with tumors that lack activating epidermal growth factor receptor (EGFR) mutations and anaplastic lymphoma kinase (ALK) fusions.

DETAILED DESCRIPTION:
Adult patients with a histologically or cytologically documented metastatic NSCLC, with tumors that lack activating EGFR mutations and ALK fusions, are eligible for enrollment. Patients will be randomized in a 1:1:1 ratio to receive treatment with durvalumab + tremelimumab combination therapy + SoC chemotherapy, durvalumab monotherapy + SoC chemotherapy, or SoC chemotherapy alone. Tumor evaluation scans will be performed until objective disease progression as efficacy assessment. All patients will be followed for survival until the end of the study. An independent data monitoring committee (IDMC) composed of independent experts will be convened to confirm the safety and tolerability of the proposed dose and schedule.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, patients should fulfill the following criteria:

1. Aged at least 18 years.
2. Histologically or cytologically documented Stage IV NSCLC.
3. Confirmed tumor PD-L1 status prior to randomization.
4. Patients must have tumors that lack activating EGFR mutations and ALK fusions.
5. No prior chemotherapy or any other systemic therapy for metastatic NSCLC.
6. World Health Organization (WHO)/Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. No prior exposure to immunemediated therapy, excluding therapeutic anticancer vaccines.

Exclusion Criteria:

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

1. Mixed small-cell lung cancer and NSCLC histology, sarcomatoid variant.
2. Active or prior documented autoimmune or inflammatory disorders.
3. Brain metastases or spinal cord compression unless the patient's condition is stable and off steroids.
4. Active infection including tuberculosis, hepatitis B, hepatitis C, or human immunodeficiency virus.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1186 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2027-11-15 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojin Shi, M.D., MSc, Study Director — One MedImmune Way, Gaithersburg, Maryland 20878, United States
Locations (134):
- United States (16):
  - Research Site, Phoenix, Arizona
  - Research Site, Bakersfield, California
  - Research Site, Santa Monica, California
  - Research Site, Fort Myers, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Louisville, Kentucky
  - Research Site, Kansas City, Missouri
  - Research Site, Canton, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Chattanooga, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Richmond, Virginia
- Brazil (9):
  - Research Site, Barretos
  - Research Site, Belo Horizonte
  - Research Site, Curitiba
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, Rio de Janeiro
  - Research Site, Santo André
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Bulgaria (3):
  - Research Site, Plovdiv
  - Research Site, Sofia
  - Research Site, Varna
- China (20):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Kunming
  - Research Site, Linyi
  - Research Site, Liuchow
  - Research Site, Nanjing
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shantou
  - Research Site, Wuhan
  - Research Site, Xining
  - Research Site, Yangzhou
  - Research Site, Zhanjiang
  - Research Site, Zhengzhou
- Germany (10):
  - Research Site, Berlin
  - Research Site, Essen
  - Research Site, Freiburg im Breisgau
  - Research Site, Gauting
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Immenhausen
  - Research Site, Mainz
  - Research Site, Oldenburg
  - Research Site, Würzburg
- Research Site, Shatin, Hong Kong
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Törökbálint
- Japan (17):
  - Research Site, Bunkyō City
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hiroshima
  - Research Site, Iwakuni-shi
  - Research Site, Kanazawa
  - Research Site, Kashiwa
  - Research Site, Kōtoku
  - Research Site, Kurume-shi
  - Research Site, Matsuyama
  - Research Site, Okayama
  - Research Site, Sapporo
  - Research Site, Sayama
  - Research Site, Sunto-gun
  - Research Site, Toyoake-shi
  - Research Site, Ube-shi
  - Research Site, Yokohama
- Mexico (7):
  - Research Site, Aguascalientes
  - Research Site, Cuautitlán Izcalli
  - Research Site, Guadalajara
  - Research Site, Mexico City
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Tuxtla Gutiérrez
- Peru (3):
  - Research Site, Arequipa
  - Research Site, Lima
  - Research Site, San Isidro
- Poland (4):
  - Research Site, Olsztyn
  - Research Site, Tomaszów Mazowiecki
  - Research Site, Warsaw
  - Research Site, Wodzisław Śląski
- Russia (3):
  - Research Site, Moscow
  - Research Site, Omsk
  - Research Site, Saint Petersburg
- South Africa (7):
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, Johannesburg
  - Research Site, Parktown
  - Research Site, Pretoria
  - Research Site, Rondebosch
  - Research Site, Vereeniging
- South Korea (7):
  - Research Site, Busan
  - Research Site, Chungcheongbuk-do
  - Research Site, Daegu
  - Research Site, Incheon
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Ulsan
- Taiwan (6):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (3):
  - Research Site, Bangkok
  - Research Site, Muang
  - Research Site, Songkhla
- Ukraine (9):
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kirovohrad
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Odesa
  - Research Site, Sumy
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhia
- United Kingdom (3):
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Manchester
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] He JZ, Duval V, Jauslin P, Goncalves A, Abegesah A, Fan C, Lim K, Song X, Chen C, Shi X, Mann H, Krug L, Ren S, Phipps A, Gibbs M, Zhou D. Population Pharmacokinetics and Exposure-Response Analysis for the CTLA-4 Inhibitor Tremelimumab in Metastatic NSCLC Patients in the Phase III POSEIDON Study. Clin Pharmacol Ther. 2023 Dec;114(6):1375-1386. doi: 10.1002/cpt.3063. Epub 2023 Oct 17. PMID 37777827
- [Derived] Johnson ML, Cho BC, Luft A, Alatorre-Alexander J, Geater SL, Laktionov K, Kim SW, Ursol G, Hussein M, Lim FL, Yang CT, Araujo LH, Saito H, Reinmuth N, Shi X, Poole L, Peters S, Garon EB, Mok T; POSEIDON investigators. Durvalumab With or Without Tremelimumab in Combination With Chemotherapy as First-Line Therapy for Metastatic Non-Small-Cell Lung Cancer: The Phase III POSEIDON Study. J Clin Oncol. 2023 Feb 20;41(6):1213-1227. doi: 10.1200/JCO.22.00975. Epub 2022 Nov 3. PMID 36327426
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419MC00004&attachmentIdentifier=7d96582a-99c4-430c-8f40-cb5baed12064&fileName=Redacted_-_D419MC00004_-___Statistical_Analysis_Plan.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419MC00004&attachmentIdentifier=650e89de-fa9b-4961-8f7f-dc89fc9ca2f5&fileName=Redacted_-_D419MC00004-csp-v6.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419MC00004&attachmentIdentifier=b9aa2703-787f-44a6-a44f-681aadf21610&fileName=Redacted_-_D419MC00004_CSR_Synopsis_-clinical-study-report.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted in 142 study centers across 18 countries in North and Latin America, Europe, Asia Pacific and Africa. First patient randomized: 27 June 2017. Results are presented for the global cohort at final analysis data cut-offs (DCOs) of 24 July 2019 (Response Evaluation Criteria in Solid Tumors [RECIST]-based endpoints) and 12 March 2021 (all other data). Once global enrollment was complete, enrollment was started in mainland China. Results for the China cohort will be reported later.
Pre-assignment Details: Patients were randomized in a stratified manner as per programmed cell death ligand 1 (PD-L1) tumor expression status (PD-L1 tumor cells [TC] ≥50% versus [vs] <50%), disease stage (IVA vs IVB), and histology (non-squamous vs squamous) in a 1:1:1 ratio to receive treatment with tremelimumab + durvalumab combination therapy + standard of care (SoC) chemotherapy (also referred to as T+ D + SoC), durvalumab monotherapy + SoC chemotherapy (also referred to as D + SoC), or SoC chemotherapy alone.
Groups:
- T + D + SoC: During chemotherapy (combination) stage:
  Patients received tremelimumab 75 milligrams (mg) + durvalumab 1500 mg combination therapy + SoC chemotherapy via intravenous (IV) infusion every 3 weeks (Q3W) for 4 doses/cycles (Weeks 0, 3, 6 and 9).
  The SoC chemotherapy was the Investigator's choice of one of the following regimens: abraxane + carboplatin (squamous and non-squamous patients), pemetrexed + cisplatin or carboplatin (non-squamous patients only), or gemcitabine + cisplatin or carboplatin (squamous patients only).
  Post-chemotherapy (maintenance) stage:
  Patients then continued to receive durvalumab monotherapy 1500 mg IV infusion every 4 weeks (Q4W) from Week 12 until progressive disease (PD), unless there was unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met. Patients also received an additional dose of tremelimumab 75 mg (in combination with durvalumab) at Week 16 post-chemotherapy.
  Non-squamous patients who received pemetrexed + carboplatin/cisplatin during chemotherapy stage could receive pemetrexed maintenance therapy, given Q4W from Week 12 until PD, unless contraindicated per the Investigator.
- D + SoC: During chemotherapy (combination) stage:
  Patients received durvalumab 1500 mg monotherapy + SoC chemotherapy via IV infusion Q3W for 4 doses/cycles (Weeks 0, 3, 6 and 9).
  The SoC chemotherapy was the Investigator's choice of one of the following regimens: abraxane + carboplatin (squamous and non-squamous patients), pemetrexed + cisplatin or carboplatin (non-squamous patients only), or gemcitabine + cisplatin or carboplatin (squamous patients only).
  Post-chemotherapy (maintenance) stage:
  Patients then continued to receive durvalumab monotherapy 1500 mg IV infusion Q4W from Week 12 until PD, unless there was unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met.
  Non-squamous patients who received pemetrexed + carboplatin/cisplatin during chemotherapy stage could receive pemetrexed maintenance therapy, given Q4W from Week 12 until PD, unless contraindicated per the Investigator.
- SoC Alone: During chemotherapy (combination) stage:
  Patients received SoC chemotherapy alone via IV infusion Q3W for 4 doses/cycles (Weeks 0, 3, 6 and 9). Patients could also receive SoC chemotherapy for an additional 2 cycles Q3W on Weeks 12 and 15 if clinically indicated and at the Investigator's discretion before the patient entered follow-up.
  The SoC chemotherapy was the Investigator's choice of one of the following regimens: abraxane + carboplatin (squamous and non-squamous patients), pemetrexed + cisplatin or carboplatin (non-squamous patients only), or gemcitabine + cisplatin or carboplatin (squamous patients only).
  Post-chemotherapy (maintenance) stage:
  Non-squamous patients who received pemetrexed + carboplatin/cisplatin during chemotherapy stage could receive pemetrexed maintenance therapy, given Q3W or Q4W (dependent on Investigator decision and local standards) from Week 12 until PD, unless contraindicated per the Investigator.
Period: Overall Study
Arm/Group | T + D + SoC | D + SoC | SoC Alone
Started (Randomized and included in global cohort analysis) | 338 | 338 | 337
Received Treatment | 331 | 335 | 331
Completed (Completed study or ongoing in study at primary completion date (global cohort final analysis DCO of 12 March 2021)) | 80 | 65 | 40
Not Completed | 258 | 273 | 297
Not completed — Death | 250 | 264 | 279
Not completed — Lost to Follow-up | 2 | 2 | 2
Not completed — Withdrawal by Subject | 6 | 7 | 16

BASELINE CHARACTERISTICS:
Population: Global cohort: All patients in the full analysis set (FAS), which included all randomized patients, were included in the baseline analysis. Patients were included in the analysis in the treatment arm to which they were randomized, regardless of the treatment they received.
Groups:
- T + D + SoC: During chemotherapy (combination) stage:
  Patients received tremelimumab 75 mg + durvalumab 1500 mg combination therapy + SoC chemotherapy via IV infusion Q3W for 4 doses/cycles (Weeks 0, 3, 6 and 9).
  The SoC chemotherapy was the Investigator's choice of one of the following regimens: abraxane + carboplatin (squamous and non-squamous patients), pemetrexed + cisplatin or carboplatin (non-squamous patients only), or gemcitabine + cisplatin or carboplatin (squamous patients only).
  Post-chemotherapy (maintenance) stage:
  Patients then continued to receive durvalumab monotherapy 1500 mg IV infusion Q4W from Week 12 until PD, unless there was unacceptable toxicity, withdrawal of consent, or another discontinuation criterion was met. Patients also received an additional dose of tremelimumab 75 mg (in combination with durvalumab) at Week 16 post-chemotherapy.
  Non-squamous patients who received pemetrexed + carboplatin/cisplatin during chemotherapy stage could receive pemetrexed maintenance therapy, given Q4W from Week 12 until PD, unless contraindicated per the Investigator.
- Total: Total of all reporting groups
Arm/Group | T + D + SoC | D + SoC | SoC Alone | Total
Number analyzed (Participants) | 338 | 338 | 337 | 1013
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (9.43) | 63.5 (9.10) | 63.1 (9.87) | 63.1 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 85 | 89 | 243
  Male | 269 | 253 | 248 | 770
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 205 | 182 | 179 | 566
  Black or African American | 8 | 4 | 8 | 20
  Asian | 99 | 123 | 128 | 350
  Native Hawaiian or other Pacific Islander | 2 | 0 | 0 | 2
  American Indian or Alaska Native | 12 | 17 | 9 | 38
  Other | 12 | 12 | 13 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 51 | 54 | 55 | 160
  Not Hispanic or Latino | 287 | 284 | 282 | 853
Age Categorical [Count of Participants; unit: Participants]
  ≥18 to <50 | 29 | 27 | 30 | 86
  ≥50 to <65 | 162 | 142 | 146 | 450
  ≥65 to <75 | 112 | 130 | 121 | 363
  ≥75 | 35 | 39 | 40 | 114

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS); D + SoC Compared With SoC Alone
Description: PFS (per RECIST version 1.1 [RECIST 1.1] using Blinded Independent Central Review [BICR] assessments) was defined as time from date of randomization until date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the patient withdrew from randomized therapy or received another anticancer therapy prior to progression. Median PFS was calculated using the Kaplan-Meier technique. The final analysis of PFS in the global cohort was pre-specified after approximately 497 BICR PFS events occurred across the D + SoC and SoC alone treatment arms (75% maturity).
Time Frame: Tumor scans performed at baseline, Week 6, Week 12 and then every 8 weeks relative to date of randomization until radiological progression. Assessed until global cohort DCO of 24 July 2019 (maximum of approximately 25 months).
Population: Global cohort: The FAS included all randomized patients. Analysis of PFS was assessed as a primary outcome measure for comparison of the D + SoC vs SoC alone treatment arms only. The alternative treatment arm comparisons were assessed as a secondary outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | D + SoC | SoC Alone
Number analyzed (Participants) | 338 | 337
months | 5.5 [4.7 to 6.5] | 4.8 [4.6 to 5.8]
Statistical Analysis 1: Comparison: D + SoC vs SoC Alone; D + SoC vs SoC alone. A hazard ratio (HR) <1 favors D + SoC to be associated with a longer PFS than SoC alone; Test type: Superiority; p = 0.00093, Log Rank — Analysis was performed using a stratified log-rank test adjusting for PD-L1 tumor expression (TC ≥50% vs <50%), histology (squamous vs non-squamous) and disease stage (IVA vs IVB) and using the Breslow approach for handling ties; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.620 to 0.885] — The HR and confidence interval (CI) were estimated from a stratified Cox proportional hazards model adjusting for PD-L1 (TC ≥50% vs <50%), histology (squamous vs non-squamous) and disease stage (IVA vs IVB) and using Efron method to control for ties

2. Primary Outcome: Overall Survival (OS); D + SoC Compared With SoC Alone
Description: OS was defined as the time from the date of randomization until death due to any cause. Any patient not known to have died at the time of analysis was censored based on the last recorded date on which the patient was known to be alive. Median OS was calculated using the Kaplan-Meier technique. The final analysis of OS in the global cohort was pre-specified after approximately 532 OS events occurred across the D + SoC and SoC alone treatment arms (80% maturity).
Time Frame: From baseline until death due to any cause. Assessed until global cohort DCO of 12 March 2021 (maximum of approximately 45 months).
Population: Global cohort: The FAS included all randomized patients. Analysis of OS was assessed as a primary outcome measure for comparison of the D + SoC vs SoC alone treatment arms only. The alternative treatment arm comparisons were assessed as a secondary outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | D + SoC | SoC Alone
Number analyzed (Participants) | 338 | 337
months | 13.3 [11.4 to 14.7] | 11.7 [10.5 to 13.1]
Statistical Analysis 1: Comparison: D + SoC vs SoC Alone; D + SoC vs SoC alone. An HR <1 favors D + SoC to be associated with a longer OS than SoC alone; Test type: Superiority; p = 0.07581, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.724 to 1.016] — The HR and CI were estimated from a stratified Cox proportional hazards model adjusting for PD-L1 (TC ≥50% vs <50%), histology (squamous vs non-squamous) and disease stage (IVA vs IVB) and using Efron method to control for ties

3. Secondary Outcome: PFS; T + D + SoC Compared With SoC Alone and T + D + SoC Compared With D + SoC
Description: PFS (per RECIST 1.1 using BICR assessments) was defined as time from date of randomization until date of objective disease progression or death (by any cause in the absence of progression), regardless of whether the patient withdrew from randomized therapy or received another anticancer therapy prior to progression. Median PFS was calculated using the Kaplan-Meier technique.
Time Frame: Tumor scans performed at baseline, Week 6, Week 12 and then every 8 weeks relative to date of randomization until radiological progression. Assessed until global cohort DCO of 24 July 2019 (maximum of approximately 25 months.
Population: Global cohort: The FAS included all randomized patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | T + D + SoC | D + SoC | SoC Alone
Number analyzed (Participants) | 338 | 338 | 337
months | 6.2 [5.0 to 6.5] | 5.5 [4.7 to 6.5] | 4.8 [4.6 to 5.8]
Statistical Analysis 1: Comparison: T + D + SoC vs SoC Alone; T + D + SoC vs SoC alone. An HR <1 favors T + D + SoC to be associated with a longer PFS than SoC alone; Test type: Superiority; p = 0.00031, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.600 to 0.860] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: OS; T + D + SoC Compared With SoC Alone and T + D + SoC Compared With D + SoC
Description: OS was defined as the time from the date of randomization until death due to any cause. Any patient not known to have died at the time of analysis was censored based on the last recorded date on which the patient was known to be alive. Median OS was calculated using the Kaplan-Meier technique.
Time Frame: as for outcome 2
Population: Global cohort: The FAS included all randomized patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | T + D + SoC | D + SoC | SoC Alone
Number analyzed (Participants) | 338 | 338 | 337
months | 14.0 [11.7 to 16.1] | 13.3 [11.4 to 14.7] | 11.7 [10.5 to 13.1]
Statistical Analysis 1: Comparison: T + D + SoC vs SoC Alone; T + D + SoC vs SoC alone. An HR <1 favors T + D + SoC to be associated with a longer OS than SoC alone; Test type: Superiority; p = 0.00304, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.650 to 0.916] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR (per RECIST 1.1 using BICR assessments) was defined as the percentage of patients with at least one visit response of complete response (CR) or partial response (PR). Results are presented for the pre-specified ORR analysis using unconfirmed responses based on BICR.
Time Frame: as for outcome 1
Population: Global cohort: The FAS included all randomized patients. The denominator was a subset of the FAS who had measurable disease at baseline.
Measure: Number; unit: percentage of patients
Arm/Group | T + D + SoC | D + SoC | SoC Alone
Number analyzed (Participants) | 335 | 330 | 332
percentage of patients | 46.3 | 48.5 | 33.4
Statistical Analysis 1: Comparison: D + SoC vs SoC Alone; D + SoC vs SoC alone. An odds ratio >1 favors D + SoC compared to SoC alone. Analysis was performed using logistic regression adjusting for PD-L1 tumor expression (TC ≥50% vs <50%), histology (squamous vs non-squamous) and disease stage (IVA vs IVB), with the CI calculated using a profile likelihood approach; Test type: Superiority; Odds Ratio (OR) = 1.90, 95% CI 2-sided [1.382 to 2.619]
Statistical Analysis 2: Comparison: T + D + SoC vs SoC Alone; T + D + SoC vs SoC alone. An odds ratio >1 favors T + D + SoC compared to SoC alone. Analysis was performed using logistic regression adjusting for PD-L1 tumor expression (TC ≥50% vs TC <50%), histology (squamous vs non-squamous) and disease stage (IVA vs IVB), with the CI calculated using a profile likelihood approach; Test type: Superiority; Odds Ratio (OR) = 1.72, 95% CI 2-sided [1.260 to 2.367]

6. Secondary Outcome: Best Objective Response (BoR)
Description: The BoR was calculated based on the overall visit responses from each RECIST 1.1 assessment. BOR was defined as the best response a patient had following randomization, but prior to starting any subsequent cancer therapy and up to and including RECIST 1.1 progression or the last evaluable assessment in the absence of RECIST 1.1 progression, as determined by BICR. Categorization of BoR was based on RECIST using the following 'response' categories: CR and PR and the following 'non-response' categories: stable disease (SD) ≥6 weeks, progression (ie, PD) and not evaluable (NE). Results are presented for number (%) of patients in each specified category.
Time Frame: as for outcome 1
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | T + D + SoC | D + SoC | SoC Alone
Number analyzed (Participants) | 335 | 330 | 332
Participants
  CR | 2 | 3 | 0
  PR | 153 | 157 | 111
  SD ≥6 weeks | 120 | 107 | 150
  PD | 48 | 60 | 61
  NE | 12 | 3 | 10

7. Secondary Outcome: Duration of Response (DoR)
Description: DoR (per RECIST 1.1 using BICR assessments) was defined as the time from the date of first documented response until date of documented progression or death in the absence of disease progression. The end of response coincided with the date of progression or death from any cause used for the RECIST 1.1 PFS endpoint. The time of the initial response was defined as the latest of the dates contributing towards the first visit of PR or CR. Results are presented for the pre-specified DoR analysis using unconfirmed responses based on BICR.
Time Frame: as for outcome 1
Population: Global cohort: The FAS included all randomized patients. Only patients with an objective response were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | T + D + SoC | D + SoC | SoC Alone
Number analyzed (Participants) | 155 | 160 | 111
months | 7.4 [3.5 to NA] — 75th percentile could not be calculated as it was not reached. | 6.0 [3.4 to NA] — 75th percentile could not be calculated as it was not reached. | 4.2 [3.0 to 6.9]

8. Secondary Outcome: Time From Randomization to Second Progression (PFS2)
Description: PFS2 was defined as the time from the date of randomization to the earliest of the progression event (subsequent to that used for the primary variable PFS) or death. The date of second progression was recorded by the Investigator and defined according to local standard clinical practice and could involve any of: objective radiological imaging, symptomatic progression or death.
Time Frame: as for outcome 1
Population: Global cohort: The FAS included all randomized patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | T + D + SoC | D + SoC | SoC Alone
Number analyzed (Participants) | 338 | 338 | 337
months | 10.4 [9.4 to 12.2] | 10.2 [9.0 to 11.5] | 9.4 [8.6 to 10.4]
Statistical Analysis 1: Comparison: D + SoC vs SoC Alone; D + SoC vs SoC alone. An HR <1 favors D + SoC to be associated with a longer PFS2 than SoC alone; Test type: Superiority; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.666 to 0.928] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: T + D + SoC vs SoC Alone; T + D + SoC vs SoC alone. An HR <1 favors T + D + SoC to be associated with a longer PFS2 than SoC alone; Test type: Superiority; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.632 to 0.883] — [estimate comment as in outcome 2, analysis 1]

9. Secondary Outcome: Pharmacokinetics (PK) of Durvalumab; Peak and Trough Serum Concentrations
Description: To evaluate PK, blood samples were collected at pre-specified timepoints and peak and trough serum concentrations of durvalumab were determined. Peak concentration on Week 0 is the post-infusion concentration of Week 0 (collected within 10 minutes of the end of infusion). Trough concentrations on Weeks 3 and 12 are the pre-infusion concentrations of Weeks 3 and 12, respectively.
Time Frame: Samples were collected post-dose on Day 1 (Week 0), pre-dose on Weeks 3 and 12 and at follow-up (3 months after the last valid dose). Assessed at the global cohort DCO of 12 March 2021.
Population: Global cohort: The PK analysis set included all patients who received at least 1 dose of durvalumab or tremelimumab per the protocol for whom any post-dose PK data were available and without any protocol deviations that would significantly affect the PK analyses. PK for durvalumab was performed for the T + D + SoC and D + SoC treatment arms only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (μg/mL)
Arm/Group | T + D + SoC | D + SoC
Number analyzed (Participants) | 327 | 330
micrograms/milliliter (μg/mL)
  Week 0: number analyzed (Participants) | 286 | 303
  Week 0 | 418.80 (164.20) | 505.01 (48.76)
  Week 3: number analyzed (Participants) | 284 | 285
  Week 3 | 82.08 (84.38) | 91.53 (100.58)
  Week 12: number analyzed (Participants) | 218 | 226
  Week 12 | 195.62 (58.65) | 212.11 (60.37)
  Follow-up (3 months): number analyzed (Participants) | 59 | 53
  Follow-up (3 months) | 13.42 (166.36) | 16.06 (249.88)

10. Secondary Outcome: PK of Tremelimumab; Peak and Trough Serum Concentrations
Description: To evaluate PK, blood samples were collected at pre-specified timepoints and peak and trough serum concentrations of tremelimumab were determined. Peak concentration on Week 0 is the post-infusion concentration of Week 0 (collected within 10 minutes of the end of infusion). Trough concentrations on Weeks 3 and 12 are the pre-infusion concentrations of Weeks 3 and 12, respectively.
Time Frame: as for outcome 9
Population: Global cohort: The PK analysis set included all patients who received at least 1 dose of durvalumab or tremelimumab per the protocol for whom any post-dose PK data were available and without any protocol deviations that would significantly affect the PK analyses. PK for tremelimumab was performed for the T + D + SoC treatment arm only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | T + D + SoC
Number analyzed (Participants) | 327
μg/mL
  Week 0: number analyzed (Participants) | 294
  Week 0 | 23.17 (65.62)
  Week 3: number analyzed (Participants) | 285
  Week 3 | 4.16 (80.83)
  Week 12: number analyzed (Participants) | 183
  Week 12 | 7.82 (75.68)
  Follow-up (3 months): number analyzed (Participants) | 105
  Follow-up (3 months) | 0.86 (87.65)

11. Secondary Outcome: Number of Patients With Anti-Drug Antibody (ADA) Response to Durvalumab
Description: Blood samples were collected at pre-specified timepoints and number of patients who developed detectable ADAs against durvalumab was determined. ADA prevalence is defined as percentage of patients with positive ADA result at any time, baseline or post-baseline. Treatment-emergent ADA is defined as either treatment-induced ADA or treatment-boosted ADA. ADA incidence is percentage of patients who were treatment-emergent ADA-positive. Treatment-boosted ADA is defined as baseline positive ADA titer that was boosted by ≥4-fold during the study period. Persistently positive is defined as having ≥2 post-baseline ADA positive measurements with ≥16 weeks (112 days) between the first and last positive, or an ADA positive result at the last available assessment. Transiently positive is defined as having ≥1 post-baseline ADA positive measurement and not fulfilling the conditions for persistently positive. Presence of neutralizing antibody (nAb) was tested for all ADA positive samples.
Time Frame: Samples were collected on Day 1 (Week 0), Week 12 and at 3 months after the last dose of study treatment (ie, durvalumab).
Population: Global cohort: The ADA evaluable patients included those in the safety analysis set with non-missing baseline ADA sample and at least 1 post-baseline ADA sample. ADA for durvalumab was performed for the T + D + SoC and D + SoC treatment arms only. The denominator was durvalumab ADA evaluable patients.
Measure: Count of Participants; unit: Participants
Arm/Group | T + D + SoC | D + SoC
Number analyzed (Participants) | 286 | 285
Participants
  ADA positive at any visit (ADA prevalence) | 42 | 33
  Treatment-emergent ADA positive (ADA incidence) | 29 | 19
  Treatment-boosted ADA | 2 | 1
  Treatment-induced ADA (ADA positive post-baseline only) | 27 | 18
  ADA positive at baseline only | 8 | 13
  ADA positive post-baseline and positive at baseline | 7 | 2
  Persistently positive | 8 | 7
  Transiently positive | 26 | 13
  nAb positive at any visit | 3 | 3

12. Secondary Outcome: Number of Patients With ADA Response to Tremelimumab
Description: Blood samples were collected at pre-specified timepoints and number of patients who developed detectable ADAs against tremelimumab was determined. ADA prevalence is defined as percentage of patients with positive ADA result at any time, baseline or post-baseline. Treatment-emergent ADA is defined as either treatment-induced ADA or treatment-boosted ADA. ADA incidence is percentage of patients who were treatment-emergent ADA-positive. Treatment-boosted ADA is defined as baseline positive ADA titer that was boosted by ≥4-fold during the study period. Persistently positive is defined as having ≥2 post-baseline ADA positive measurements with ≥16 weeks (112 days) between the first and last positive, or an ADA positive result at the last available assessment. Transiently positive is defined as having ≥1 post-baseline ADA positive measurement and not fulfilling the conditions for persistently positive. Presence of nAb was tested for all ADA positive samples.
Time Frame: Samples were collected on Day 1 (Week 0), Week 12 and at 3 months after the last dose of study treatment (ie, tremelimumab).
Population: Global cohort: The ADA evaluable patients included those in the safety analysis set with non-missing baseline ADA sample and at least 1 post-baseline ADA sample. ADA for tremelimumab was performed for the T + D + SoC treatment arm only. The denominator was tremelimumab ADA evaluable patients.
Measure: Count of Participants; unit: Participants
Arm/Group | T + D + SoC
Number analyzed (Participants) | 278
Participants
  ADA positive at any visit (ADA prevalence) | 44
  Treatment-emergent ADA positive (ADA incidence) | 38
  Treatment-boosted ADA | 3
  Treatment-induced ADA (ADA positive post-baseline only) | 35
  ADA positive at baseline only | 4
  ADA positive post-baseline and positive at baseline | 5
  Persistently positive | 22
  Transiently positive | 18
  nAb positive at any visit | 31

13. Secondary Outcome: Time to Deterioration of Global Health Status / Health-Related Quality of Life (HRQoL) and Patient Reported Outcome (PRO) Symptoms, Assessed Using European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)
Description: The EORTC QLQ-Core 30 version 3 (QLQ-C30 v3) was included for assessing HRQoL. It assesses HRQoL/health status through 9 multi-item scales: 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, and nausea and vomiting), and a global health and QoL scale. 6 single-item symptom measures are also included: dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties. Scores from 0 to 100 were derived for each of the 15 domains, with higher scores representing greater functioning, greater HRQoL, or greater level of symptoms. Time to deterioration was defined as time from randomization until the date of first clinically meaningful deterioration that was confirmed at a subsequent visit or death (by any cause) in the absence of a clinically meaningful deterioration.
Time Frame: At baseline, Weeks 3, 6, 9, 12, 16 and 20, then Q4W until PD, on Day 28 and 2 months post-PD, then every 8 weeks until second progression/death (whichever came first). Assessed until global cohort DCO of 12 March 2021 (maximum of approximately 45 months).
Population: Global cohort: The FAS included all randomized patients. For QLQ-C30 function scales and global health status/HRQoL, only patients with baseline scores ≥10 (and with data available) were included in the analysis. For QLQ-C30 symptom scales/items, only patients with baseline scores ≤90 (and with data available) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | T + D + SoC | D + SoC | SoC Alone
Number analyzed (Participants) | 325 | 326 | 321
months
  QLQ-C30 Global Health Status / HRQoL: number analyzed (Participants) | 319 | 321 | 318
  QLQ-C30 Global Health Status / HRQoL | 8.3 [6.4 to 10.2] | 7.8 [6.5 to 9.5] | 5.6 [4.4 to 7.5]
  QLQ-C30 Physical Functioning: number analyzed (Participants) | 323 | 325 | 320
  QLQ-C30 Physical Functioning | 7.7 [5.9 to 9.4] | 8.3 [6.6 to 10.0] | 5.3 [4.2 to 6.5]
  QLQ-C30 Role Functioning: number analyzed (Participants) | 314 | 313 | 304
  QLQ-C30 Role Functioning | 6.6 [5.4 to 8.3] | 7.4 [5.8 to 9.3] | 4.8 [3.6 to 6.2]
  QLQ-C30 Cognitive Functioning: number analyzed (Participants) | 323 | 323 | 318
  QLQ-C30 Cognitive Functioning | 7.6 [6.1 to 9.7] | 7.4 [5.6 to 9.3] | 5.8 [4.6 to 7.5]
  QLQ-C30 Emotional Functioning: number analyzed (Participants) | 322 | 322 | 315
  QLQ-C30 Emotional Functioning | 8.5 [6.6 to 11.3] | 9.5 [7.4 to 12.0] | 7.5 [5.8 to 11.0]
  QLQ-C30 Social Functioning: number analyzed (Participants) | 320 | 319 | 314
  QLQ-C30 Social Functioning | 6.4 [5.6 to 9.4] | 7.1 [5.0 to 9.6] | 5.7 [4.6 to 7.4]
  QLQ-C30 Fatigue: number analyzed (Participants) | 317 | 318 | 314
  QLQ-C30 Fatigue | 3.7 [2.8 to 5.0] | 3.8 [2.9 to 4.9] | 2.8 [2.1 to 3.7]
  QLQ-C30 Pain: number analyzed (Participants) | 316 | 311 | 298
  QLQ-C30 Pain | 8.9 [6.2 to 10.9] | 6.5 [5.6 to 8.6] | 5.7 [4.6 to 7.2]
  QLQ-C30 Nausea / Vomiting: number analyzed (Participants) | 322 | 322 | 319
  QLQ-C30 Nausea / Vomiting | 7.8 [5.6 to 10.0] | 5.6 [4.1 to 6.6] | 5.6 [4.2 to 7.5]
  QLQ-C30 Dyspnea: number analyzed (Participants) | 310 | 310 | 301
  QLQ-C30 Dyspnea | 7.9 [5.8 to 9.8] | 6.9 [5.8 to 8.9] | 6.7 [5.5 to 8.8]
  QLQ-C30 Insomnia: number analyzed (Participants) | 311 | 304 | 301
  QLQ-C30 Insomnia | 8.3 [6.4 to 10.4] | 7.4 [5.6 to 9.8] | 5.8 [4.2 to 7.2]
  QLQ-C30 Appetite Loss: number analyzed (Participants) | 308 | 316 | 305
  QLQ-C30 Appetite Loss | 7.2 [5.7 to 9.4] | 7.2 [4.7 to 8.8] | 7.0 [5.6 to 9.6]
  QLQ-C30 Constipation: number analyzed (Participants) | 315 | 314 | 306
  QLQ-C30 Constipation | 9.2 [6.4 to 12.2] | 8.7 [6.5 to 10.0] | 6.1 [4.8 to 7.5]
  QLQ-C30 Diarrhea: number analyzed (Participants) | 324 | 324 | 320
  QLQ-C30 Diarrhea | 11.0 [9.3 to 13.6] | 9.8 [8.1 to 12.9] | 10.8 [9.2 to 15.1]

14. Secondary Outcome: Time to Deterioration of PRO Symptoms, Assessed Using EORTC QLQ-Lung Cancer Module 13 (QLQ-LC13)
Description: The EORTC QLQ-LC13 is a disease-specific 13-item self-administered questionnaire for lung cancer, to be used in conjunction with the EORTC QLQ-C30. It comprises both multi-item and single-item measures of lung cancer-associated symptoms (ie, coughing, hemoptysis, dyspnea, and pain) and treatment-related symptoms from conventional chemotherapy and radiotherapy (ie, hair loss, neuropathy, sore mouth, and dysphagia). Scores from 0 to 100 were derived for each symptom item, with higher scores representing greater level of symptoms. Time to deterioration was defined as time from randomization until the date of first clinically meaningful deterioration that was confirmed at a subsequent visit or death (by any cause) in the absence of a clinically meaningful deterioration.
Time Frame: as for outcome 13
Population: Global cohort: The FAS included all randomized patients. For QLQ-LC13 symptom scales/items, only patients with baseline scores ≤90 (and with data available) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | T + D + SoC | D + SoC | SoC Alone
Number analyzed (Participants) | 325 | 326 | 321
months
  QLQ-LC13 Cough: number analyzed (Participants) | 302 | 314 | 295
  QLQ-LC13 Cough | 9.7 [7.3 to 13.3] | 11.0 [8.7 to 13.5] | 8.8 [6.8 to 12.3]
  QLQ-LC13 Hemoptysis: number analyzed (Participants) | 325 | 326 | 318
  QLQ-LC13 Hemoptysis | 17.8 [12.5 to 31.3] | 14.0 [10.3 to 21.4] | 11.4 [9.3 to 19.3]
  QLQ-LC13 Dyspnea: number analyzed (Participants) | 325 | 325 | 316
  QLQ-LC13 Dyspnea | 5.4 [4.2 to 6.4] | 5.0 [3.8 to 6.4] | 3.6 [2.6 to 4.5]
  QLQ-LC13 Pain in Chest: number analyzed (Participants) | 319 | 322 | 309
  QLQ-LC13 Pain in Chest | 10.0 [7.7 to 13.3] | 9.5 [7.8 to 11.8] | 8.6 [6.8 to 11.4]
  QLQ-LC13 Pain in Arm or Shoulder: number analyzed (Participants) | 312 | 311 | 310
  QLQ-LC13 Pain in Arm or Shoulder | 8.9 [6.6 to 10.9] | 8.9 [7.4 to 10.3] | 8.8 [6.2 to 12.0]
  QLQ-LC13 Pain in Other Parts: number analyzed (Participants) | 312 | 314 | 306
  QLQ-LC13 Pain in Other Parts | 9.7 [6.8 to 12.1] | 8.9 [6.8 to 11.2] | 5.8 [4.9 to 9.3]

ADVERSE EVENTS:
Time Frame: Adverse events: from first dose of study treatment until the earlier of 90 days after last dose or the date of first subsequent anticancer therapy. All-cause mortality (death due to any cause): from randomization up to global cohort final analysis DCO (12 March 2021). Maximum timeframe of approximately 45 months.
Description: Safety analysis set included all patients who received at least 1 dose of study treatment (analyzed according to actual treatment received). 1 patient randomized to T + D + SoC arm and 1 patient randomized to D + SoC arm only received SoC and were included in SoC alone arm of the safety analysis set. All-cause mortality was determined for patients in the FAS (analyzed according to randomized treatment arm, regardless of the treatment received). Results are reported for the global cohort only.
Arm/Group | T + D + SoC | D + SoC | SoC Alone
All-Cause Mortality (participants affected / at risk) | 251/338 | 265/338 | 285/337
Serious Adverse Events (participants affected / at risk) | 146/330 | 134/334 | 117/333
Other Adverse Events (participants affected / at risk) | 309/330 | 302/334 | 301/333
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T + D + SoC (N=330) | D + SoC (N=334) | SoC Alone (N=333)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Autoimmune pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 5 (5) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 3 (4) | 2 (2)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (2) | 2 (2)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 18 (32) | 23 (30) | 21 (25)
Neutropenia (Blood and lymphatic system disorders) | 4 (5) | 6 (8) | 3 (5)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 2 (2) | 2 (2)
Cardiac death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 5 (6) | 3 (4)
Death (General disorders) | 3 (3) | 6 (6) | 1 (1)
Face oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (2) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 8 (8) | 1 (1) | 1 (1)
Sudden death (General disorders) | 1 (1) | 3 (3) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (8) | 6 (7) | 3 (3)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 3 (3) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Abscess oral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute hepatitis B (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 3 (3) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Candida pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 3 (4)
Chikungunya virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Encephalitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Nosocomial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Autoimmune myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 36 (42) | 21 (23) | 16 (17)
Pneumonia bacterial (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 3 (4) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 5 (5) | 2 (2) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0) | 3 (3)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 3 (6)
Platelet count decreased (Investigations) | 2 (2) | 2 (2) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Mandibular mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Polymyositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cancer fatigue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0)
Eyelid naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 3 (3) | 2 (2) | 3 (4)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 4 (4) | 1 (1) | 1 (1)
Coordination abnormal (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalitis autoimmune (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Polyneuropathy in malignant disease (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Spinal cord disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Device occlusion (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Deafness bilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 4 (4) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Autoimmune nephritis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Bladder mass (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 3 (3) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 5 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 7 (8) | 3 (3)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 9 (9)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 3 (3)
Diabetes insipidus (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (7) | 5 (5) | 4 (4)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 2 (2) | 1 (1) | 0 (0)
Brachiocephalic vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T + D + SoC (N=330) | D + SoC (N=334) | SoC Alone (N=333)
Abdominal pain (Gastrointestinal disorders) | 19 (22) | 16 (19) | 10 (10)
Constipation (Gastrointestinal disorders) | 63 (85) | 72 (98) | 79 (96)
Diarrhoea (Gastrointestinal disorders) | 65 (98) | 57 (72) | 49 (66)
Leukopenia (Blood and lymphatic system disorders) | 41 (80) | 32 (59) | 39 (80)
Nausea (Gastrointestinal disorders) | 136 (281) | 120 (258) | 121 (243)
Anaemia (Blood and lymphatic system disorders) | 150 (213) | 137 (188) | 146 (203)
Neutropenia (Blood and lymphatic system disorders) | 98 (177) | 75 (135) | 77 (161)
Stomatitis (Gastrointestinal disorders) | 17 (18) | 20 (25) | 16 (17)
Vomiting (Gastrointestinal disorders) | 59 (82) | 51 (74) | 45 (80)
Asthenia (General disorders) | 56 (67) | 31 (42) | 39 (49)
Fatigue (General disorders) | 81 (116) | 80 (119) | 74 (93)
Mucosal inflammation (General disorders) | 17 (19) | 11 (15) | 6 (6)
Oedema peripheral (General disorders) | 27 (35) | 23 (29) | 30 (34)
Pyrexia (General disorders) | 48 (65) | 30 (38) | 22 (30)
Thrombocytopenia (Blood and lymphatic system disorders) | 56 (83) | 38 (67) | 54 (77)
Upper respiratory tract infection (Infections and infestations) | 22 (32) | 12 (13) | 18 (27)
Alanine aminotransferase increased (Investigations) | 45 (66) | 43 (63) | 44 (59)
Amylase increased (Investigations) | 28 (47) | 24 (41) | 16 (27)
Aspartate aminotransferase increased (Investigations) | 42 (67) | 36 (59) | 38 (51)
Blood creatinine increased (Investigations) | 21 (33) | 12 (16) | 12 (21)
Gamma-glutamyltransferase increased (Investigations) | 18 (18) | 17 (20) | 11 (11)
Lipase increased (Investigations) | 20 (34) | 12 (23) | 7 (12)
Neutrophil count decreased (Investigations) | 39 (66) | 46 (96) | 59 (110)
Platelet count decreased (Investigations) | 22 (28) | 19 (24) | 29 (35)
Weight decreased (Investigations) | 23 (23) | 29 (30) | 20 (24)
White blood cell count decreased (Investigations) | 24 (44) | 21 (50) | 27 (53)
Decreased appetite (Metabolism and nutrition disorders) | 92 (115) | 71 (89) | 81 (117)
Hyperglycaemia (Metabolism and nutrition disorders) | 18 (28) | 18 (25) | 12 (13)
Hypokalaemia (Metabolism and nutrition disorders) | 25 (38) | 11 (19) | 14 (20)
Hyponatraemia (Metabolism and nutrition disorders) | 9 (12) | 16 (19) | 18 (25)
Arthralgia (Musculoskeletal and connective tissue disorders) | 41 (55) | 28 (31) | 20 (23)
Back pain (Musculoskeletal and connective tissue disorders) | 25 (27) | 16 (21) | 15 (16)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 18 (21) | 9 (9) | 20 (20)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 (20) | 8 (9) | 8 (8)
Dizziness (Nervous system disorders) | 20 (22) | 22 (28) | 9 (15)
Headache (Nervous system disorders) | 37 (49) | 23 (29) | 24 (26)
Insomnia (Psychiatric disorders) | 26 (30) | 40 (42) | 29 (36)
Cough (Respiratory, thoracic and mediastinal disorders) | 33 (39) | 38 (42) | 22 (23)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30 (30) | 29 (32) | 24 (25)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 16 (22) | 17 (24)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 19 (20) | 9 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 33 (34) | 36 (38) | 20 (20)
Hyperthyroidism (Endocrine disorders) | 19 (20) | 20 (21) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 36 (43) | 30 (41) | 15 (18)
Rash (Skin and subcutaneous tissue disorders) | 63 (81) | 46 (58) | 22 (23)
Hypothyroidism (Endocrine disorders) | 39 (42) | 21 (24) | 4 (4)
Hypertension (Vascular disorders) | 20 (21) | 9 (13) | 6 (9)

LIMITATIONS AND CAVEATS:
This study also incorporates a China tail, comprising additional patients randomized after the end of the global cohort recruitment. Efficacy and safety of patients randomized in China will be reported at a later date once this separate analysis has been completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/16/NCT03164616/Prot_002.pdf
  • Statistical Analysis Plan (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/16/NCT03164616/SAP_003.pdf